CLINICAL TRIAL: NCT00390299
Title: Phase I Trial of a Measles Virus Derivative Producing CEA (MV-CEA) in Patients With Recurrent Glioblastoma Multiforme (GBM)
Brief Title: Viral Therapy in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC0671; NCI-2009-01198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0671 (Other: Mayo Clinic); P30CA015083 (NIH); P50CA108961 (NIH)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-01

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Mixed Glioma; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (resection cavity administration) (Experimental): Patients undergo en block resection of their tumor (after confirming diagnosis) on day 1, followed by MV-CEA administered into the resection cavity.
  Interventions: Biological: Carcinoembryonic Antigen-Expressing Measles Virus; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery
- Arm B (intratumoral and resection cavity administration) (Experimental): Patients undergo stereotactic biopsy (to confirm the diagnosis) and placement of a catheter within the tumor, followed by MV-CEA IT through the catheter over 10 minutes on day 1. Patients then undergo en block resection of their tumor with computer-assisted stereotactic techniques on day 5, followed by MV-CEA administered around the tumor bed.
  Interventions: Biological: Carcinoembryonic Antigen-Expressing Measles Virus; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Carcinoembryonic Antigen-Expressing Measles Virus — Given via injection into resection cavity or around tumor bed and/or IT
  Other Names: MV-CEA
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo en bloc resection

SUMMARY:
This phase I trial studies the side effects and best dose of carcinoembryonic antigen-expressing measles virus (MV-CEA) in treating patients with glioblastoma multiforme that has come back. A virus, called MV-CEA, which has been changed in a certain way, may be able to kill tumor cells without damaging normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and toxicity of intratumoral and resection cavity administration of an Edmonston's strain measles virus genetically engineered to produce CEA (MV-CEA) in patients with recurrent glioblastoma multiforme.

II. To determine the maximum tolerated dose (MTD) of MV-CEA. III. To characterize viral gene expression at each dose level as manifested by CEA titers.

IV. To assess viremia, viral replication, and measles virus shedding/persistence following intratumoral administration.

V. To assess humoral and cellular immune response to the injected virus. VI. To assess in a preliminary fashion antitumor efficacy of this approach.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 sequential treatment arms.

ARM A (RESECTION CAVITY ADMINISTRATION): Patients undergo en block resection of their tumor (after confirming diagnosis) on day 1, followed by MV-CEA administered into the resection cavity.

ARM B (INTRATUMORAL AND RESECTION CAVITY ADMINISTRATION): Patients undergo stereotactic biopsy (to confirm the diagnosis) and placement of a catheter within the tumor, followed by carcinoembryonic antigen-expressing measles virus intratumorally (IT) through the catheter over 10 minutes on day 1. Patients then undergo en block resection of their tumor with computer-assisted stereotactic techniques on day 5, followed by MV-CEA administered around the tumor bed.

After completion of study treatment, patients are followed up at 28 days (non-cohort I patients), 7 weeks (patients in cohort I only), every 2 months until progression, every 3 and 12 months after progression, and then yearly thereafter for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent grade 3 or 4 glioma, including astrocytoma, oligodendroglioma or mixed glioma with histologic confirmation at initial diagnosis or recurrence
* Candidate for gross total or subtotal resection
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets (PLT) >= 100,000/uL
* Total bilirubin =< 1.5 x upper normal limit (ULN)
* Aspartate aminotransferase (AST) =< 2 x ULN
* Creatinine =< 2.0 x ULN
* Hemoglobin (Hgb) >= 9.0 gm/dL
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.3 x ULN
* Ability to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Anti-measles virus immunity as demonstrated by immunoglobulin G (IgG) anti-measles antibody levels of >= 1.1 EU/ml as determined by enzyme immunoassay
* Normal serum CEA levels (< 3 ng/ml) at the time of registration
* Willing to provide biologic specimens as required by the protocol
* Negative serum pregnancy test done =< 7 days prior to registration (for women of childbearing potential only)

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Active infection =< 5 days prior to registration
* History of tuberculosis or history of purified protein derivative (PPD) positivity
* Any of the following therapies:

  * Chemotherapy =< 4 weeks prior to registration (6 wks for nitrosourea-based chemotherapy)
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Bevacizumab =< 12 weeks prior to registration
  * Non-cytotoxic antitumor drugs, i.e., small molecule cell cycle inhibitors =< 2 weeks prior to registration
  * Radiation therapy =< 6 weeks prior to registration
  * Any viral or gene therapy prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Requiring blood product support
* Inadequate seizure control
* Expected communication between ventricles and resection cavity as a result of surgery
* Human immunodeficiency virus (HIV)-positive test result, or history of other immunodeficiency
* History of organ transplantation
* History of chronic hepatitis B or C
* Other concurrent chemotherapy, immunotherapy, radiotherapy or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10-23 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Resection Cavity) - Dose Level 1: Patients undergo en block resection of their tumor (after confirming diagnosis) followed by 10^5 TCID50 MV-CEA administered into the resection cavity on day 1.
- Arm A (Resection Cavity) - Dose Level 2: Patients undergo en block resection of their tumor (after confirming diagnosis) followed by 10^6 TCID50 MV-CEA administered into the resection cavity on day 1.
- Arm A (Resection Cavity) - Dose Level 3: Patients undergo en block resection of their tumor (after confirming diagnosis) followed by 10^7 TCID50 MV-CEA administered into the resection cavity on day 1.
- Arm B (Intratumoral/Resection Cavity) - Dose Level 1: Patients undergo stereotactic biopsy (to confirm the diagnosis) and placement of a catheter within the tumor, followed by intratumoral administration of 10^6 TCID50 MV-CEA on day 1. Patients then undergo en block resection of their tumor with computer-assisted stereotactic techniques followed by injection of 10^6 TCID50 MV-CEA in resection cavity on day 5.
- Arm B (Intratumoral/Resection Cavity) - Dose Level 2: Patients undergo stereotactic biopsy (to confirm the diagnosis) and placement of a catheter within the tumor, followed by intratumoral administration of 10^7 TCID50 MV-CEA on day 1. Patients then undergo en block resection of their tumor with computer-assisted stereotactic techniques followed by injection of 10^7 TCID50 MV-CEA in resection cavity on day 5.
Period: Overall Study
Arm/Group | Arm A (Resection Cavity) - Dose Level 1 | Arm A (Resection Cavity) - Dose Level 2 | Arm A (Resection Cavity) - Dose Level 3 | Arm B (Intratumoral/Resection Cavity) - Dose Level 1 | Arm B (Intratumoral/Resection Cavity) - Dose Level 2
Started | 4 | 3 | 3 | 3 | 10
Completed | 3 | 3 | 3 | 3 | 10
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Cancellation | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Resection Cavity) - Dose Level 1 | Arm A (Resection Cavity) - Dose Level 2 | Arm A (Resection Cavity) - Dose Level 3 | Arm B (Intratumoral/Resection Cavity) - Dose Level 1 | Arm B (Intratumoral/Resection Cavity) - Dose Level 2 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 10 | 23
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <40 years | 1 | 0 | 0 | 0 | 1 | 2
  Age Group: 40-60 years | 3 | 2 | 3 | 2 | 5 | 15
  Age Group: >60 years | 0 | 1 | 0 | 1 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 8 | 11
  Male | 4 | 2 | 2 | 2 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 3 | 10 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 1 | 1 | 1 | 0 | 3 | 6
    1 | 3 | 1 | 2 | 2 | 6 | 14
    2 | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Participants With Dose-Limiting Toxicity Events (Phase I) Maximum Tolerated Dose (MTD) (Phase I) as Measured by the Number of Participants With Dose Limiting Toxicities
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Dose-limiting toxicities include hematologic events grade 3 or higher (except grade 3 ANC lasting < 72 hours), non-hematologic events graded 3 or higher (except grade 3 nausea, vomiting, or diarrhea were to be considered DLT only if patient was receiving the max supportive care and alopecia was not considered dose limiting), neurologic toxicity grade 2 or higher, grade 2 allergic reactions asymptomatic bronchospasm and/or urticarial, grade 3 or higher allergic reactions, viremia lasting for 6 weeks or more from last viral administration deemed at least possibly related to treatment. The number of patients reporting a dose-limiting event are reported.
Time Frame: 2 weeks
Population: Excludes cancel patient (never started treatment).
Measure: Number; unit: patients
Arm/Group | Arm A (Resection Cavity) - Dose Level 1 | Arm A (Resection Cavity) - Dose Level 2 | Arm A (Resection Cavity) - Dose Level 3 | Arm B (Intratumoral/Resection Cavity) - Dose Level 1 | Arm B (Intratumoral/Resection Cavity) - Dose Level 2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10
patients | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Arm A (Resection Cavity) - Dose Level 1 vs Arm A (Resection Cavity) - Dose Level 2 vs Arm A (Resection Cavity) - Dose Level 3; Test type: Other; Maximum Tolerated Dose (x 10^7 TCID50) = 1
Statistical Analysis 2: Comparison: Arm B (Intratumoral/Resection Cavity) - Dose Level 1 vs Arm B (Intratumoral/Resection Cavity) - Dose Level 2; Test type: Other; Maximum Tolerated Dose (x 10^7 TCID50) = 1

2. Primary Outcome: Number of Patients Experiencing Grade 3+ Adverse Events, Per NCI CTCAE Version 3.0
Description: The number of patients experiencing grade 3+ adverse events (overall and by arm) will be tabulated and summarized in this patient population.
Time Frame: Up to 2 weeks
Population: Per protocol analysis population; excludes cancel patient (never started treatment). Per section 16.2 of the protocol, this analysis will be performed by arm (for Arms A and B).
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Resection Cavity Administration): Patients undergo en block resection of their tumor (after confirming diagnosis) followed by MV-CEA administered into the resection cavity on day 1.
- Arm B (Intratumoral and Resection Cavity Administration): Patients undergo stereotactic biopsy (to confirm the diagnosis) and placement of a catheter within the tumor, followed by intratumoral administration of MV-CEA on day 1. Patients then undergo en block resection of their tumor with computer-assisted stereotactic techniques followed by injection of MV-CEA in resection cavity on day 5.
Arm/Group | Arm A (Resection Cavity Administration) | Arm B (Intratumoral and Resection Cavity Administration)
Number analyzed (Participants) | 9 | 13
Participants | 6 | 5

3. Secondary Outcome: Best Response, Defined as the Best Objective Status Recorded From the Start of the Treatment Until Disease Progression/Recurrence
Description: The number of responses will be summarized by simple descriptive summary statistics delineating response type. CR = total disappearance of all tumor with patient off corticosteroids or only on adrenal replacement maintenance. PR= 50% reduction in product of perpendicular diameters of contrast enhancement or mass with no new lesions with the patient being on stable or decreased steroid dose. REGR = unequivocal reduction in size of contrast-enhancement or decrease in mass effect as agreed upon independently by primary physician and quality control physicians; no new lesions. SD = failure to qualify for CR, PR, REGR, or PROG. PROG = >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions and/or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions.
Time Frame: Up to 2 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Resection Cavity Administration) | Arm B (Intratumoral and Resection Cavity Administration)
Number analyzed (Participants) | 9 | 13
Participants
  SD | 8 | 12
  PD | 1 | 1

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Percentage of patients who are progression free at 3 and 6 months (PFS3 and PFS6) will be summarized descriptively. Progression-free survival is defined as the length of time from date of registration to a) date of progression or death due to any cause or b) last follow-up. Progression is defined as a >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions, and/or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions.
Time Frame: Length of time from date of registration to a) date of progression or death due to any cause or b) last follow-up, assessed up to 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Resection Cavity Administration) | Arm B (Intratumoral and Resection Cavity Administration)
Number analyzed (Participants) | 9 | 13
percentage of patients
  PFS at 3 months | 55.6 [31.0 to 99.7] | 61.5 [40.0 to 94.6]
  PFS at 6 months | 22.2 [6.6 to 75.4] | 23.1 [8.6 to 62.3]

5. Secondary Outcome: Survival
Description: Overall survival is defined as the length of time from date of registration to a) death due to any cause or b) last follow-up. Reported using standard Kaplan-Meier estimation method.
Time Frame: Up to 13 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Resection Cavity Administration) | Arm B (Intratumoral and Resection Cavity Administration)
Number analyzed (Participants) | 9 | 13
months | 11.8 [4.4 to NA] — The 95% confidence interval upper limit was not reached. | 11.4 [4.3 to NA] — The 95% confidence interval upper limit was not reached.
Statistical Analysis 1: Comparison: Arm A (Resection Cavity Administration) vs Arm B (Intratumoral and Resection Cavity Administration); Test type: Superiority; p = 0.28, Log Rank; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.67 to 4.11]

6. Other Pre Specified Outcome: CEA Titers
Description: Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlates between these laboratory values and other outcome measures like response and dose levels will be carried out in an exploratory manner.
Time Frame: Up to 15 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in CD4 Counts
Description: as for outcome 6
Time Frame: Baseline to day 28
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in CD46 Status
Description: as for outcome 6
Time Frame: Baseline to up to day 5
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in CD8 Counts
Description: as for outcome 6
Time Frame: Baseline to day 28
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Viral Shedding
Description: as for outcome 6
Time Frame: Baseline to day 28
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Viremia
Description: as for outcome 6
Time Frame: Baseline to up to 15 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Measles Virus Specific Immunity, in Terms of Change in Interferon Gamma
Description: as for outcome 6
Time Frame: Baseline to day 28
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Measles Virus Specific Immunity, in Terms of Change in Lymphoproliferative Assay Results
Description: as for outcome 6
Time Frame: Baseline to day 28
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Viral Propagation in Tumor
Description: as for outcome 6
Time Frame: Up to day 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Description: All patients who received treatment were assessed at the end of two weeks for adverse events.
Arm/Group | Arm A (Resection Cavity) - Dose Level 1 | Arm A (Resection Cavity) - Dose Level 2 | Arm A (Resection Cavity) - Dose Level 3 | Arm B (Intratumoral/Resection Cavity) - Dose Level 1 | Arm B (Intratumoral/Resection Cavity) - Dose Level 2
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 10/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Resection Cavity) - Dose Level 1 (N=3) | Arm A (Resection Cavity) - Dose Level 2 (N=3) | Arm A (Resection Cavity) - Dose Level 3 (N=3) | Arm B (Intratumoral/Resection Cavity) - Dose Level 1 (N=3) | Arm B (Intratumoral/Resection Cavity) - Dose Level 2 (N=10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 2 (2) | 3 (6) | 8 (12)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1) | 2 (6) | 3 (3) | 7 (17)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 4 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 2 (6) | 1 (2) | 1 (1) | 1 (3) | 1 (3)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 2 (4) | 1 (1) | 4 (7)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6) | 2 (3) | 1 (1) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Seizure (Nervous system disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Speech disorder (Nervous system disorders) | 1 (1) | 1 (3) | 1 (3) | 2 (2) | 3 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT00390299/Prot_SAP_000.pdf